CLINICAL TRIAL: NCT00747032
Title: Multi-Center, Double-Blind, Randomized, Vehicle-controlled, Parallel-Group Study Comparing NYC-0462 Ointment To a Vehicle Control
Brief Title: To Demonstrate the Superior Efficacy of NYC 0462 Ointment Over That of the Placebo in the Treatment of Plaque Psoriasis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study withdrawn due to business decisions. No subjects were treated.
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Kathleen Ocasio, Nycomed US Inc.
Organization: Nycomed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYC 0462-01-01
Record Dates: First submitted 2008-09-01; First posted 2008-09-04 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): NYC 0462 Ointment
  Interventions: Drug: NYC 0462 Ointment
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NYC 0462 Ointment — To assess the efficacy of NYC 0462 Ointment versus Placebo in the treatment of Plaque Psoriasis
  Arms: 1
Drug: Placebo — To assess the efficacy of NYC 0462 Ointment versus Placebo in the treatment of Plaque Psoriasis
  Arms: 2

SUMMARY:
The aim of this trial is to assess the efficacy of NYC-0462 Ointment in the Treatment of Plaque Psoriasis.Treatment medication will be administered as follows: A thin layer of study product will be applied to the affected skin, excluding the face, once daily, at approximately the same time daily.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable, symptomatic plaque psoriasis
* Good health with the exception of psoriasis
* % BSA and plaque elevation requirements

Exclusion Criteria:

* Subjects who are pregnant, nursing or planning a pregnancy within the study participation period.
* Subjects who have any systemic or dermatological disorders with the exception of psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in plaque elevation score | 8 weeks

SECONDARY OUTCOMES:
Reduction in Investigator´s Global Evaluation, erythema and scaling scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ocasio, Study Chair — Fougera Pharmaceuticals Inc.